CLINICAL TRIAL: NCT02689258
Title: A Phase 2, Randomized, Controlled Evaluation of the Efficacy and Safety of HTX-011 or HTX-002 for Post-Operative Analgesia Following Abdominoplasty Surgery
Brief Title: Evaluation of the Efficacy and Safety of HTX-011 for Postoperative Analgesia Following Abdominoplasty Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heron Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HTX-011-C2015-203
Record Dates: First submitted 2016-02-16; First posted 2016-02-23 (Estimated); Results first posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (12):
- Part A, Cohort A: HTX-011A (Experimental): HTX- 011A (bupivacaine/meloxicam), 200 mg/6 mg via injection
  Interventions: Drug: HTX-011A
- Parts A and B, Cohort B: Saline Placebo (Placebo Comparator): Saline placebo via injection
  Interventions: Drug: Placebo
- Part A, Cohort C: HTX-011B (Experimental): HTX- 011B (bupivacaine/meloxicam), 200 mg/6 mg via injection
  Interventions: Drug: HTX-011B
- Part A, Cohort D: HTX-011B (Experimental): HTX- 011B (bupivacaine/meloxicam), 400 mg/12 mg via injection
  Interventions: Drug: HTX-011B
- Part A, Cohort E: HTX-011B (Experimental): HTX- 011B (bupivacaine/meloxicam), 400 mg/12 mg via combination
  Interventions: Drug: HTX-011B
- Part A, Cohort F: HTX-011B (Experimental): HTX- 011B (bupivacaine/meloxicam), 600 mg/18 mg via injection
  Interventions: Drug: HTX-011B
- Part B, Cohort A: HTX-002 (Experimental): HTX-002, 400 mg via combination
  Interventions: Drug: HTX-002
- Part C, Cohort A: HTX-011B (Experimental): HTX-011B (bupivacaine/meloxicam), 400 mg/12 mg via instillation
  Interventions: Drug: HTX-011B
- Part C, Cohort B: HTX-011B (Experimental): HTX-011B (bupivacaine/meloxicam), 400 mg/12 mg via combination
  Interventions: Drug: HTX-011B
- Part C, Cohort C: HTX-011B (Experimental): HTX-011B (bupivacaine/meloxicam), 300 mg/9 mg via combination
  Interventions: Drug: HTX-011B
- Part C, Cohort D: Bupivacaine HCI (Active Comparator): Bupivacaine HCl, 100 mg via injection
  Interventions: Drug: Bupivicaine HCl
- Part C, Cohort E: Saline Placebo (Placebo Comparator): Saline placebo via injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HTX-011B — HTX- 011B (bupivacaine/meloxicam) via injection
  Arms: Part A, Cohort C: HTX-011B; Part A, Cohort D: HTX-011B; Part A, Cohort E: HTX-011B; Part A, Cohort F: HTX-011B; Part C, Cohort A: HTX-011B; Part C, Cohort B: HTX-011B; Part C, Cohort C: HTX-011B
Drug: Placebo — Saline placebo via injection
  Arms: Part C, Cohort E: Saline Placebo; Parts A and B, Cohort B: Saline Placebo
Drug: HTX-011A — HTX- 011A (bupivacaine/meloxicam) via injection
  Arms: Part A, Cohort A: HTX-011A
Drug: HTX-002 — HTX-002 via combination
  Arms: Part B, Cohort A: HTX-002
Drug: Bupivicaine HCl — Bupivacaine HCl via injection
  Arms: Part C, Cohort D: Bupivacaine HCI

SUMMARY:
A Phase 2, Randomized, Controlled Evaluation of the Efficacy and Safety of HTX-011 or HTX-002 for Post-Operative Analgesia Following Abdominoplasty Surgery

DETAILED DESCRIPTION:
This study includes multiple formulations for formulation selection of the fixed-combination product and for the factorial design assessment of the contribution of the bupivacaine component. HTX-011A is the second formulation studied (HTX-011-49). HTX-011B is the final formulation studied (HTX-011-56), which was also included in subsequent Phase 2b and Phase 3 studies. For the factorial design assessment, HTX-002, a bupivacaine-only formulation in the same HTX-011 proprietary polymer was evaluated.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be considered eligible to participate in the study:

1. Be scheduled to undergo abdominoplasty surgery that is amenable to treatment with a long acting local anesthetic as per the anesthesia protocol
2. Be American Society of Anesthesiology (ASA) physical Class I or II
3. Subjects 18 years of age or older
4. Have clinical laboratory values that are within normal limits (WNL); subjects with AST/ALT < 3 x ULN, and/or creatinine < 2 x ULN are acceptable.
5. Have a body mass index ≤ 30 kg/m2
6. Female subjects are eligible only if all of the following apply:

   * Not pregnant (female subject of child bearing potential must have a negative serum pregnancy tests at screening and negative urine pregnancy test before surgery)
   * Not lactating
   * Not planning to become pregnant during the study
   * Be surgically sterile; or at least two years post-menopausal; or have a monogamous partner who is surgically sterile; or is practicing double-barrier contraception; or practicing abstinence (must agree to use double-barrier contraception in the event of sexual activity); or using an insertable, injectable, transdermal, or combination oral contraceptive approved by the FDA for greater than 2 months prior to screening visits and commits to the use of an acceptable form of birth control for the duration of the study
7. Male subjects must be surgically sterile (biologically or surgically) or commit to the use of a reliable method of birth control for the duration of the study
8. Does NOT have, as determined by the investigator or the study's medical monitor, a history or clinical manifestations of significant renal, hepatic, cardiovascular, metabolic, neurologic, psychiatric, or other condition that would preclude participation in the study
9. Must be able to understand study procedures and be willing to comply and give informed consent for the conduct of all study procedures, using an IRB approved consent

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from participating in the study:

1. Have a contraindication or be allergic to any medication to be used during the trial period
2. Have another painful physical condition that, in the opinion of the investigator, may confound the assessments of post-operative pain
3. Have a history of migraine or frequent headaches, seizures, or are currently taking anticonvulsants
4. Currently taking analgesics for a chronically painful condition, or has taken long acting opioids within 3 days of surgery, or taken any opioids within 24 hours of surgery
5. Previous abdominal surgery, as determined by the investigator, that would preclude participation in the study
6. Subjects that require liposuction as part of the abdominoplasty procedure in Part A of the protocol
7. Subjects that are to have ancillary procedures performed during the abdominoplasty surgery that are unrelated to the abdominal area (breast reduction, breast augmentation, etc.)
8. Subjects unable to discontinue medications that have not been at a stable dose for at least 14 days prior to the scheduled abdominoplasty procedure and before dosing with investigational product
9. Subjects taking the following medications; anticonvulsants, sedatives (including benzodiazepines) corticosteroids (by any means of administration), nonsteroidal anti-inflammatory drugs (NSAIDS) within 24 hours of study drug dosing, morphine, monoamine oxidase inhibitors (MAOIs), tricyclic antidepressants (TCAs), neuroleptics, or serotonin-norepinephrine reuptake inhibitors (SNRIs). Gabapentin and pregabalin are not permitted
10. Have a known or suspected history of alcohol or drug abuse
11. Have positive results on the alcohol breath test indicative of alcohol abuse or urine drug screen indicative of illicit drug use (unless results can be explained by a current prescription or acceptable over-the-counter medication at screening as determined by the investigator). The urine drug screen prior to surgery must be negative
12. Have evidence of a clinically significant 12-lead ECG abnormality according to the judgment of the investigator
13. Have received any investigational product within 30 days before start of study
14. Have previously received HTX-011 in clinical trials
15. Experiences a clinically significant event during surgery prior to the administration of the investigational product (e.g., excessive bleeding, hemodynamic instability) that would render the subject medically unstable, complicate their post-surgical course, or significantly increase the risk of study drug administration as per the judgment of the investigator. This will result in the subject being reported as randomized, not treated.
16. Subjects with sleep apnea or are on home continuous positive airway pressure (CPAP)
17. Subjects who are receiving oxygen therapy at the time of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2016-02-23 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Phoenix, Arizona
  - Pasadena, California
  - Pasadena, Maryland
  - Bellaire, Texas
  - Houston, Texas
  - Plano, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 Subject underwent complete abdominoplasty and was unintentionally randomized to receive HTX-002 (intended for mini-abdominoplasty procedure only). This subject is included in the Safety, ITT, and mITT Populations.
Groups:
- Part C, Cohort D: Bupivacaine HCI: Bupivacaine HCl 100 mg via injection.
Period: Overall Study
Arm/Group | Part A, Cohort A: HTX-011A | Parts A and B, Cohort B: Saline Placebo | Part A, Cohort C: HTX-011B | Part A, Cohort D: HTX-011B | Part A, Cohort E: HTX-011B | Part A, Cohort F: HTX-011B | Part B, Cohort A: HTX-002 | Part C, Cohort A: HTX-011B | Part C, Cohort B: HTX-011B | Part C, Cohort C: HTX-011B | Part C, Cohort D: Bupivacaine HCI | Part C, Cohort E: Saline Placebo
Started | 20 | 63 | 10 | 11 | 17 | 10 | 17 | 17 | 27 | 35 | 17 | 32
Completed | 20 | 59 | 10 | 11 | 16 | 10 | 17 | 17 | 25 | 35 | 17 | 31
Not Completed | 0 | 4 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Not completed — Subject Non-Compliance | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Subject Refusal to Continue | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Other | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study HTX-011-203 included multiple study parts, various study drugs, formulations, and administration techniques. It was pre-specified in the SAP to pool different doses of the same study drug within study parts for Participant Flow, Baseline Characteristics, and AEs. We pooled different doses of the same study drug within study parts for Participant Flow, Baseline Characteristics, and AEs. However for Outcome Measures, different doses of study drugs were presented separately.
Groups:
- Part A, Cohorts C Through F: HTX-011B: Cohort C: HTX- 011B (bupivacaine/meloxicam), 200 mg/6 mg via injection; Cohort D: HTX- 011B (bupivacaine/meloxicam), 400 mg/12 mg via injection; Cohort E: HTX- 011B (bupivacaine/meloxicam), 400 mg/12 mg via combination; Cohort F: HTX- 011B (bupivacaine/meloxicam), 600 mg/18 mg via injection.
- Part C, Cohort A Through C: HTX-011B: Cohort A: HTX-011B (bupivacaine/meloxicam), 400 mg/12 mg via instillation; Cohort B: HTX-011B (bupivacaine/meloxicam), 400 mg/12 mg via combination; Cohort C: HTX-011B (bupivacaine/meloxicam), 300 mg/9 mg via combination.
- Total: Total of all reporting groups
Arm/Group | Part A, Cohort A: HTX-011A | Parts A and B, Cohort B: Saline Placebo | Part A, Cohorts C Through F: HTX-011B | Part B, Cohort A: HTX-002 | Part C, Cohort A Through C: HTX-011B | Part C, Cohort D: Bupivacaine HCI | Part C, Cohort E: Saline Placebo | Total
Number analyzed (Participants) | 20 | 63 | 48 | 17 | 77 | 17 | 32 | 274
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (10.11) | 43.3 (10.56) | 41.0 (9.66) | 47.3 (9.77) | 39.9 (9.44) | 40.6 (6.38) | 43.2 (8.53) | 41.8 (9.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 63 | 46 | 17 | 77 | 17 | 32 | 272
  Male | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
  Asian | 2 | 4 | 1 | 1 | 3 | 0 | 0 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 13 | 13 | 4 | 16 | 4 | 9 | 64
  White | 13 | 45 | 31 | 12 | 57 | 13 | 23 | 194
  More than one race | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 63 | 48 | 17 | 77 | 17 | 32 | 274

OUTCOME MEASURES:

1. Primary Outcome: Summed Pain Intensity Scores Collected Over 24 Hours
Description: The SPI is derived by summing the pain intensity score weighted by the scheduled time duration. SPI0-24 will be calculated by summing the Pain intensity (PI) score at the relevant time points weighted by the scheduled time duration since the prior PI assessment as follows: SPI0-24= PI1+PI2+2*PI4+2*PI6+2*PI8+2*PI10+2*PI12+2*PI14+4*PI18+6*PI24. Min = 0 (if PI=0 at every time) and Max = 240 (if PI=10 at every time).
Time Frame: 24 hours
Population: mITT Population.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Part A, Cohort A: HTX-011A | Parts A and B, Cohort B: Saline Placebo
Number analyzed (Participants) | 20 | 63
Units on a scale | 92.60 (47.531) | 96.16 (43.775)

2. Primary Outcome: Summed Pain Intensity Scores Collected Over 24 Hours
Description: as for outcome 1
Time Frame: 24 Hours
Population: mITT Population.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Part A, Cohort C: HTX-011B | Part A, Cohort D: HTX-011B | Part A, Cohort E: HTX-011B | Part A, Cohort F: HTX-011B | Part B, Cohort A: HTX-002
Number analyzed (Participants) | 10 | 11 | 17 | 10 | 17
Units on a scale | 79.53 (40.458) | 74.64 (46.893) | 66.38 (53.214) | 89.46 (45.402) | 83.85 (37.326)

3. Primary Outcome: Summed Pain Intensity Scores Collected Over 24 Hours
Description: as for outcome 1
Time Frame: 24 Hours
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Part C, Cohort A: HTX-011B | Part C, Cohort B: HTX-011B | Part C, Cohort C: HTX-011B | Part C, Cohort D: Bupivacaine HCI | Part C, Cohort E: Saline Placebo
Number analyzed (Participants) | 17 | 25 | 35 | 17 | 32
Units on a scale | 113.72 (49.109) | 83.23 (43.966) | 104.65 (44.140) | 110.22 (41.980) | 121.93 (52.530)

ADVERSE EVENTS:
Time Frame: 28 Days.
Description: Study HTX-011-202 included multiple study parts, various study drugs, formulations, and administration techniques. It was pre-specified in the SAP to pool different doses of the same study drug within study parts for Participant Flow, Baseline Characteristics, and AEs. We pooled different doses of the same study drug within study parts for Participant Flow, Baseline Characteristics, and AEs. However for Outcome Measures, different doses of study drugs were presented separately.
Arm/Group | Part A, Cohort A: HTX-011A | Parts A and B, Cohort B: Saline Placebo | Part A, Cohorts C Through F: HTX-011B | Part B, Cohort A: HTX-002 | Part C, Cohort A Through C: HTX-011B | Part C, Cohort D: Bupivacaine HCI | Part C, Cohort E: Saline Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/63 | 0/48 | 0/17 | 0/77 | 0/17 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/63 | 0/48 | 0/17 | 1/77 | 1/17 | 0/32
Other Adverse Events (participants affected / at risk) | 19/20 | 50/63 | 42/48 | 13/17 | 67/77 | 15/17 | 27/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A, Cohort A: HTX-011A (N=20) | Parts A and B, Cohort B: Saline Placebo (N=63) | Part A, Cohorts C Through F: HTX-011B (N=48) | Part B, Cohort A: HTX-002 (N=17) | Part C, Cohort A Through C: HTX-011B (N=77) | Part C, Cohort D: Bupivacaine HCI (N=17) | Part C, Cohort E: Saline Placebo (N=32)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A, Cohort A: HTX-011A (N=20) | Parts A and B, Cohort B: Saline Placebo (N=63) | Part A, Cohorts C Through F: HTX-011B (N=48) | Part B, Cohort A: HTX-002 (N=17) | Part C, Cohort A Through C: HTX-011B (N=77) | Part C, Cohort D: Bupivacaine HCI (N=17) | Part C, Cohort E: Saline Placebo (N=32)
Incision site infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 0
Headache (Nervous system disorders) | 3 | 13 | 16 | 4 | 16 | 2 | 11
Dizziness (Nervous system disorders) | 3 | 8 | 5 | 3 | 4 | 4 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 3 | 0 | 1 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 2 | 0 | 1 | 1 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 2 | 0 | 3 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 2 | 2 | 1 | 0 | 7 | 2 | 0
Hypotension (Vascular disorders) | 1 | 3 | 5 | 1 | 4 | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 11 | 37 | 22 | 6 | 46 | 12 | 14
Constipation (Gastrointestinal disorders) | 8 | 9 | 15 | 3 | 24 | 7 | 10
Flatulence (Gastrointestinal disorders) | 0 | 2 | 3 | 0 | 1 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 3 | 1 | 3 | 12 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 0 | 1 | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 9 | 4 | 1 | 9 | 2 | 6
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 4 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 1 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 3 | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 6 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 2 | 2 | 0 | 1 | 1 | 1
Polyuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Labia enlarged (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 1 | 0 | 4 | 2 | 3
Chills (General disorders) | 1 | 1 | 0 | 0 | 4 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 2 | 0 | 0 | 0
Liver function test increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 3 | 2 | 2 | 10 | 2 | 4
Incision site erythema (Injury, poisoning and procedural complications) | 0 | 4 | 0 | 0 | 1 | 0 | 0
Incision site hypoaesthesia (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Incision site swelling (Injury, poisoning and procedural complications) | 0 | 4 | 0 | 0 | 0 | 0 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 5 | 0 | 3
Wound complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0 | 2
Wound secretion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 4 | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Swelling (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Incision site pruritus (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-02-06): https://cdn.clinicaltrials.gov/large-docs/58/NCT02689258/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-23): https://cdn.clinicaltrials.gov/large-docs/58/NCT02689258/SAP_001.pdf